CLINICAL TRIAL: NCT04793763
Title: Comparing the Effect of Deep Neck Flexors and MCkenice Exercises on Cervical Mobility,Pain and Disability in Chronic Neck Pain Participants
Brief Title: Comparing the Effect of Deep Neck Flexors Versus MCkenice Exercises on Cervical Functions
Acronym: McKENICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Diab, professor of physical therapy cairo university, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003053
Record Dates: First submitted 2021-02-19; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Chronic Neck Pain
Keywords: Mc Kenzie; chronic neck pain; deep neck flexor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Placebo Comparator): placebo Comparator Group A
  : twenty patients were received traditional Physical Therapy agents
  Interventions: Other: traditional therapeutic exercises
- group B (Experimental): experimental Group B Group B: twenty patients were received traditional Physical Therapy agents plus isometric, stretching, scapulothoracic exercises and deep neck flexors exercises;
  Interventions: Other: traditional therapeutic exercises and McKenize technique
- group C (Experimental): Experimental Group C
  Group C: twenty patients were received traditional Physical Therapy agents plus isometric, stretching, scapulothoracic exercises and Mckenzie technique.
  Interventions: Other: traditional therapeutic exercises and deep neck flexor exercises

INTERVENTIONS:
Other: traditional therapeutic exercises — group A will receive traditional exercises
  Arms: group A
Other: traditional therapeutic exercises and McKenize technique — Group B will receive traditional therapeutic exercises and McKenize technique
  Arms: group B
Other: traditional therapeutic exercises and deep neck flexor exercises — Group C receive traditional therapeutic exercises and deep neck flexor exercises
  Arms: group C

SUMMARY:
Physical Therapy rehabilitation programs could involve Manual procedures, stretching, traction, massage, electrotherapy, thermal agents, ultrasound, education and general exercise..In the recovery of patients with neck pain, exercise is one of the most commonly used modalities to gain muscle strength, endurance, and flexibility in order to recover damaged muscles and to maintain regular life activities.. Neck pain management exercise programs vary in terms of length, training frequency, intensity, and mode of exercise. .

DETAILED DESCRIPTION:
This study will be a randomized controlled trial that involved sixty patients of both gender with chronic neck pain with duration of at least six weeks that will be recruited into the study. They will be recruited from the out patient clinic of Faculty of Physical Therapy, Egypt ,their age ranged from (30-50) years old with mean age, their height ranged from (152-182) cm and their weight ranged from (55-90) kg , Patients will be included if they had a localized chronic neck pain without any current arm pain or discomfort were included.Groups:

A: twenty patients will receive traditional Physical Therapy agents, Group B: twenty patients will receive traditional Physical Therapy agents plus isometric, stretching, scapulothoracic exercises and deep neck flexors exercises; and Group C: twenty patients will receive traditional Physical Therapy agents plus isometric, stretching, scapulothoracic exercises and Mckenzie technique.

ELIGIBILITY:
Inclusion Criteria:

1. age ranges from (30-50) years old with mean age,
2. height ranges from (152-182) cm and their weight ranged from (55-90) kg
3. Patients will be included if they have a localized chronic neck pain without any current arm pain or discomfort were included.

Exclusion Criteria:

1. history of cervical spine injury or surgery, if neck pain is secondary to other conditions (including neoplasm, neurological diseases or vascular diseases),
2. they have a radiculopathy presenting neurological deficit
3. they had infection or inflammatory arthritis in the cervical spine,
4. they have pain with any cause in or around the scapula, shoulder, upper extremities and lumbar spine that prevents stabilization of these structures.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
neck functional activity | after 6 weeks
  The Copenhagen neck capacity inability scale
pain disability | after 6 weeks
  VAS
cervical range of motion | after 6 weeks
  use Myrin goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Abd el aziem, professor, Study Director — Cairo University
Locations (1):
- Faculity of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No